CLINICAL TRIAL: NCT03058588
Title: Next Generation Sequencing (NGS) Approach to Study Known and New Germline Mutations in Familial Acute Myeloid Leukemia and Myelodisplastic Syndromes
Brief Title: Next Generation Sequencing (NGS) in Familial Acute Myeloid Leukemia and Myelodisplastic Syndromes
Status: Recruiting | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Prof Domenico Russo, Full Professor of Hematology, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NEXT-FAMLY 1016
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor DNA of index case will be extracted from 10 ml of PB collected at diagnosis in EDTA tubes. Mononuclear cells from PB (PBMC)will be separated and isolated by Ficoll gradient. Tumor DNA will be extracted possibly soon after the isolation. Tumor DNA of affected relative/-s will be extracted from PBMC isolated at diagnosis, or during the patients monitoring, and stored at -80°C. Tumor DNA previously extracted and stored at -20°C may be used in event of no PB or bone marrow sample available.
  Germline DNA of index case and relatives will be extracted by buccal epithelial cells isolated by Isohelix SK-2 DNA Buccal Swab Collection Kit by Therapak Corporation, Isohelix SK-2 DNA Buccal Swab Collection Kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Analysis with molecular biology: Any patient with acute leukemia or other myeloid malignancy AND
  1. a first- or second-degree relative with acute leukemia or other myeloid malignancies
  2. a first- or second-degree relative with lymphoproliferative neoplasms
  3. or with clinical features that resemble one of the familial myeloid malignancies predisposition syndromes
  Interventions: Genetic: Analysis with molecular biology

INTERVENTIONS:
Genetic: Analysis with molecular biology — Molecular screening by next generation sequencing (NGS) platform, for known and unknown mutations potentially associated with the disease

SUMMARY:
The aim of this study is to look for predisposing mutations in patients and relatives affected by AML and MDS with familial history of myeloid or, less frequently, lymphoid malignancies. Taking advantage of a next generation sequencing (NGS) platform, screening for known and unknown mutations potentially associated with the disease will be done. The screening will be performed on affected and unaffected family members, in order to outline new pedigrees that either validate previous findings or constitute novel discoveries.

DETAILED DESCRIPTION:
Patients with a diagnosis of AML or MDS with at least one relative affected by AL/MDS or, secondly, lymphoproliferative disorders, will be enrolled into the study, and will be referred to as the index case. The analysis will be performed both retrospectively and prospectively. A gene panel deep sequencing (GPDS) of the tumor DNA from peripheral blood of the index case at diagnosis will be performed in order to identify mutations in a number of genes known to be associated to myeloid malignancies, mainly: ASXL1, BCOR, NRAS, TP53, RUNX1, CEBPA, FLT3, EZH2, IDH1, IDH2, NPM1, DNMT3A, TET2, CBL, KRAS, ETV6, SF3B1, SRSF2, U2AF1, ZRSR2, GATA2, TERT, TERC, SRP72, and ANKRD26.

In case none of the known mutations is found by the GPDS, whole exome sequencing (WES) will be performed as second step on the tumor cells of the index case.

When one or multiple somatic mutations are found, a Sanger Sequencing (SS) on germline DNA from epithelial buccal cells of the index cases and affected relatives will be performed for the screening of the same somatic leukemic mutations on germline DNA. If the index case and affected relatives share the same mutations on the germline, the same germline mutations will be checked by SS in the unaffected family members.

ELIGIBILITY:
Inclusion criteria:

Any patient with acute myeloid leukemia (AML) or Myelodisplastic Syndrome (MDS) with:

1. a first- or second-degree relative with Acute leukemia or MDS or other myeloid malignancies
2. a first- or second-degree relative with Lymphoproliferative neoplasms
3. or with clinical features that resemble one of the familial MDS/AML predisposition syndromes:

   * History of thrombocytopenia and/or a clinical bleeding propensity (as in RUNX1, ANKRD26 or ETV6 germline mutations)
   * Abnormal nails or skin pigmentation, oral leukoplakia, idiopathic pulmonary fibrosis, unexplained liver disease (as in TERT and TERC germline mutations)
   * Lymphedema, atypical infections, immune deficiencies (as in GATA2 germline mutations)

Exclusion Criteria:

1. any diagnosis other than acute myeloid leukemia (AML) or Myelodisplastic Syndrome (MDS);
2. acute myeloid leukemia (AML) or Myelodisplastic Syndrome (MDS) without a first- or second-degree relative with Acute leukemia or MDS or other myeloid malignancies or without a first- or second-degree relative with Lymphoproliferative neoplasms or with clinical features that resemble one of the familial MDS/AML predisposition syndromes;
3. unability to sign the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Detailed personal and family history from every patient affected by myeloid malignancy will be obtained, in order to identify patients with at least one relative affected by myeloid malignancy or lymphoproliferative disorders or with the features that increase the likelihood of one of the aforementioned familial myeloid malignancy predisposition syndromes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-02-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Discovery of predisposing mutations | After enrollment of the first 10 cases (an avarage of 2 years)
  Screening of tumor and germline DNA for predisposing mutations

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Russo, MD, Principal Investigator — Chair of Hematology
Locations (1):
- Chair of Hematology and Bone marrow Transplant Unit, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No